CLINICAL TRIAL: NCT07048912
Title: The Effect of Acute Beetroot Juice Supplementation on Anaerobic Performance in Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melike Nur Eroğlu (Other)
Responsible Party: Sponsor-Investigator, Melike Nur Eroğlu, Lecturer, Sakarya Applied Sciences University
Organization: Sakarya Applied Sciences University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: SUBU-EROGLU-2025-01
Record Dates: First submitted 2025-06-11; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Exercise Performance; Supplementation
Keywords: beetroot juice; muscle oxygenation; nitrate; football; high intensity efforts

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot Juice (BJ) (Experimental): Participants in this arm consumed 140 mL of nitrate-rich beetroot juice (~12.8 mmol nitrate) as a single acute dose, approximately 2.5 hours before the performance assessments. The supplementation was administered in the morning under supervision, and participants were instructed to maintain their usual diet but avoid additional nitrate-rich foods 24 hours prior to testing.
  Interventions: Dietary Supplement: Beetroot Juice (BJ); Dietary Supplement: Blackcurrant Juice (Placebo)
- Placebo (Experimental): Participants in this arm consumed 140 mL of blackcurrant juice containing negligible nitrate (<0.1 mmol) as a single acute dose, approximately 2.5 hours before the performance assessments. The supplementation was administered in the morning under supervision, and participants followed the same dietary instructions as the experimental group, avoiding nitrate-rich foods 24 hours prior to testing.
  Interventions: Dietary Supplement: Beetroot Juice (BJ); Dietary Supplement: Blackcurrant Juice (Placebo)

INTERVENTIONS:
Dietary Supplement: Beetroot Juice (BJ) — This intervention involves a single 140 mL dose of a commercially available concentrated beetroot juice supplement (Beet-It Pro Elite Shot, James White Drinks Ltd., UK), containing approximately 12.8 mmol (800 mg) of dietary nitrate. Participants consume the juice 2.5 hours prior to performing a 30-second Wingate anaerobic test. The purpose of this intervention is to examine its acute effects on anaerobic performance, muscle oxygenation, and metabolic responses.
Dietary Supplement: Blackcurrant Juice (Placebo) — This intervention involves a single 140 mL dose of a low-calorie blackcurrant juice (Pfanner, Austria) with negligible nitrate content (<0.1 mmol). The placebo is matched to beetroot juice in appearance, taste, and packaging to ensure double-blind conditions. It is consumed 2.5 hours before the Wingate test and serves as the control condition.

SUMMARY:
The aim of this clinical trial is to examine the effects of two different natural fruit-vegetable blend beverages on short-duration, high-intensity exercise performance and muscle oxygenation in young male football players. The study also investigates how these beverages influence certain metabolic responses. The main questions it seeks to answer are:

* Does one of the beverages improve peak and mean power output during the Wingate test?
* How do these beverages affect muscle oxygenation and post-exercise recovery?
* Researchers will compare the effects of the two beverages on performance and metabolic markers.

Participants:

* Consume one of the two natural beverages 2.5 hours before testing (assigned at random)
* Perform a 30-second high-intensity Wingate cycling test
* Undergo measurements of muscle oxygenation, heart rate, blood pressure, blood lactate, and blood glucose during and after exercise
* Maintain consistent dietary and physical activity routines and avoid certain foods prior to testing

ELIGIBILITY:
Inclusion Criteria:

* Healthy males over 18 years old
* Performing resistance exercise at least three times per week
* At least 5 years of football training experience

Exclusion Criteria:

* Contraindications to Wingate exercise
* Presence of cardiometabolic disease
* Current use of ergogenic supplementation
* Smokers

Ages: 18 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Mean power output during the 30-second Wingate anaerobic test | Day 1 (2.5 hours after supplementation, during Wingate test)
  Average power (in watts) generated during the 30-second Wingate cycling test will be compared between beetroot juice and placebo conditions to assess anaerobic performance.

SECONDARY OUTCOMES:
Muscle oxygen saturation (SmO₂) | Day 1 (pre-, during, and post-exercise on the day of Wingate test)
  SmO₂ will be assessed using Near-Infrared Spectroscopy (NIRS) on the vastus lateralis muscle. Measurements will be taken continuously before, during, and after the 30-second Wingate anaerobic test to evaluate changes in muscle oxygenation in response to the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University of Applied Sciences, Faculty of Sport Sciences, Exercise and Sports Sciences Education, Application and Research Centre, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We prefer not to share the Individual Participant Data (IPD) to protect participant privacy and comply with data protection and ethical guidelines.

DOCUMENTS (1):
  • Informed Consent Form (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT07048912/ICF_000.pdf